CLINICAL TRIAL: NCT00740064
Title: A Pilot Study of Highly Active Antiretroviral Therapy Using Isentress (Raltegravir) and Epzicom (Abacavir/Lamivudine) in Antiretroviral Naive HIV-Infected Subjects
Brief Title: Pilot Study With Isentress (Raltegravir) and Epzicom (Abacavir/Lamivudine) in Treatment Naive HIV-Infected Subjects
Acronym: SHIELD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Denver Infectious Disease Consultants, PLLC (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Benjamin Young, MD, PhD, Denver Infectious Disease Consultants, PLLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COL111429
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: HIV Infections
Keywords: HIV infections
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; abacavir; Lamivudine; abacavir, lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Raltegravir and Abacavir/Lamivudine — Raltegravir 400mg BID Abacavir/Lamivudine 1 tablet QD
  Other Names: Isentress; Epzicom; RTG; ABC/3TC

SUMMARY:
To evaluate the efficacy and safety of Raltegravir and Epzicom over 48 weeks in ART-naive HIV-infected subjects.

DETAILED DESCRIPTION:
* This is a single-arm, multicenter, open-label, pilot study to evaluate the efficacy, safety, and tolerability of RTG BID and ABC/3TC QD. A total of 30 subjects will be enrolled at 3 U.S. sites.
* The study includes a 30-day screening period, a treatment period (baseline through week 48), and a follow-up visit, 2 to 4 weeks after the last study visit, as needed to resolve any ongoing AEs or to confirm virologic status.

Virologic failure (VF) is defined as having either virologic non-response or virologic rebound. Virologic failure is confirmed by having 2 consecutive plasma HIV-1 RNA levels taken at least 2 weeks apart according to the following definitions:

* virologic rebound is defined as HIV-1 RNA level ≥400 copies/mL after initial response of HIV-1 RNA <400 copies/mL or >1 log10 copies/mL increase above nadir;
* virologic non-response is defined as HIV-1 RNA >400 copies/mL at week 24.
* Subjects will be discontinued from the study if virologic failure is confirmed. When a subject is suspected to have virologic failure, a confirmatory HIV-1 RNA must be performed at an unscheduled visit between 2 weeks and 4 weeks after the initial assessment, and a plasma sample collected for resistance testing.
* Subjects who experience symptoms consistent with a clinically suspected ABC HSR must permanently discontinue ABC/3TC, and will be allowed to substitute study-provided fixed-dose combination ZDV/3TC 150/300 mg (COMBIVIR®) BID for ABC/3TC and remain in the study.

ELIGIBILITY:
Inclusion Criteria:

* Antiretroviral naïve defined as ≤7 days of ART prior to study entry
* Negative for HLA-B*5701 allele
* Screening HIV-1 RNA >1,000 copies/mL
* Screening laboratory values:

  * Hemoglobin > 8.0 g/dL
  * Platelet count >50,000/mm3
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase <5 x ULN
  * Total bilirubin <2.5 x ULN
  * Absolute neutrophil count >500/mm3
  * Calculated creatinine clearance (CrCL) ≥50 mL/min by Cockcroft-Gault:
  * For men, (140 - age in years) x (body weight in kg) ÷ (serum creatinine in mg/dL x 72) = CrCl (mL/min)*
  * For women, multiply the result by 0.85 = CrCl (mL/min)
* A female subject is eligible to participate in the study if she is of:
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal); or,
* Childbearing potential with a negative pregnancy test at screen and agrees to use one of the following methods of contraception (any contraception method must be used consistently and correctly, i.e., in accordance with both the product label and the instructions of a physician):
* Agreement for complete abstinence from intercourse from 2 weeks prior to administration of investigational products, throughout the study, and for 2 weeks after discontinuation of all study medications.
* Double barrier contraception (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide);
* Any intrauterine device (IUD) with published data showing that the expected failure rate is less than 1% per year (not all IUDs meet this criterion);
* Any other method with published data showing that the lowest expected failure rate for the method is less than 1% per year.
* Men and women age (≥18 years).
* Ability and willingness of subject to give written informed consent.

Exclusion Criteria:

* Screening HIV-1 genotype indicating the presence of any of the following mutations: K65R, L74V, and Y115F or a combination of two or more thymidine analog mutations (M41L, D67N, K70R, K219Q or E) that include changes at either L210 or T215, associated with ABC and 3TC resistance, and mutations Q148H/R/K and N155H associated with RTG resistance.
* Currently pregnant or breast-feeding.
* Hepatitis B infection with chronic viral replication (HBsAg+).
* Presence of a serious medical condition, including but not limited to congestive heart failure, cardiomyopathy or other cardiac dysfunction, which in the opinion of the investigator would compromise the safety of the subject.
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry. NOTE: Use of corticosteroids for acute therapy for PCP is permitted. Prednisone at a daily dose of 10 mg or less (physiologic replacement dose) or short course corticosteroid therapy (≤ 10 days) is permitted.
* Known allergy/sensitivity to study drugs or their formulations.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Illnesses that are determined serious by the site investigator, (i.e. requiring systemic treatment and/or hospitalization) until subject either completes therapy or is clinically stable on therapy, for at least 7 days prior to study entry.
* Requirement for medications that are not allowed to be taken with study treatment.
* Current imprisonment or involuntary incarceration in a medical facility for psychiatric or physical (e.g. infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-08 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy and safety of RTG and ABC/3TC over 48 weeks in ART-naive HIV-infected subjects. | 48 weeks

SECONDARY OUTCOMES:
To assess the immunologic response, changes in fasting lipids, renal function, and development of resistance of the study regimen | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Young, MD, PhD, Principal Investigator — Denver Infectious Disease Consultants, PLLC
Locations (3):
- United States (3):
  - Spectrum Medical Group, Phoenix, Arizona
  - Denver Infectious Disease Consultants, PLLC, Denver, Colorado
  - Southwest CARE Center, Santa Fe, New Mexico